CLINICAL TRIAL: NCT03005028
Title: Angiogram Based Fractional Flow Reserve FFRangio - A Validation Study
Status: Completed | Type: Observational
Sponsor: CathWorks Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: FFRAngio 1.0
Record Dates: First submitted 2016-12-19; First posted 2016-12-29 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: CAD - Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Control

SUMMARY:
In the present study we aim at validating the computation of FFRangio values from the angiogram by comparing them to measured wire-based FFR values, in a larger scale and in a completely blinded manner. Investigation of a wide range of users in various conditions may strengthen the reliability of the FFRAngio measurements.

ELIGIBILITY:
Inclusion Criteria:

* Male and female above 18 years old age which undergo FFR as part of their standard care
* TIMI Grade Flow is equal to 3
* LVEF larger than 45%.
* Subjects with multi-vessel coronary artery disease, with NSTEMI are allowed.

Exclusion Criteria:

* Contraindicated for FFR examination or adenosine administration
* STEMI
* CTO
* TIMI Grade Flow below 3
* Arteries supplying akinetic or severe hypokinetic territories
* Prior CABG on the study vessel
* Left Main stenosis, In-stent restenosis and Collaterals
* Diffused atherosclerosis diseases and tandem lesions
* Aorto-ostial lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll male and female subjects above the age of 18, with stable angina who were referred to coronary angiography and have an FFR measurement in at least one coronary artery.
Sampling Method: Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03-15 (Actual); Study Completion 2016-03-15 (Actual)

PRIMARY OUTCOMES:
Lesion-specific image-based FFRAngio calculation, compared to the invasive FFR as the reference gold standard, with a blinded analysis yielding Bland- Altman of +/- 15% with 95% CI | 1 hour
  Immediately following the invasive FFR procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pellicano M, Lavi I, De Bruyne B, Vaknin-Assa H, Assali A, Valtzer O, Lotringer Y, Weisz G, Almagor Y, Xaplanteris P, Kirtane AJ, Codner P, Leon MB, Kornowski R. Validation Study of Image-Based Fractional Flow Reserve During Coronary Angiography. Circ Cardiovasc Interv. 2017 Sep;10(9):e005259. doi: 10.1161/CIRCINTERVENTIONS.116.005259. PMID 28916602